CLINICAL TRIAL: NCT00545584
Title: Multicenter, Open, Pragmatic, Randomized Trial Comparing the Efficacy of 3 Different Lifestyle Interventions After Addition of Sitagliptin to Patients With Type 2 Diabetes Mellitus Who Have Inadequate Glycemic Control on Metformin Therapy
Brief Title: Addition Of Januvia (Sitagliptin) Improves Glycemic Control In Patients Inadequately Controlled By Metformin (MK0431-078)
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 0431-078; 2007_023
Record Dates: First submitted 2007-10-16; First posted 2007-10-17 (Estimated); Results first posted 2011-05-11 (Estimated); Last update posted 2017-05-12 (Actual); Status verified 2017-04

CONDITIONS: Diabetes Mellitus, Non-Insulin-Dependent
MeSH Terms: conditions — Diabetes Mellitus, Type 2 | interventions — Sitagliptin Phosphate

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Sitagliptin with Standard of Care (Experimental): Subjects received sitagliptin 100 mg once daily for 26 Weeks, and: No specific intervention (standard recommendation) on physical exercise and diet.
  Interventions: Drug: sitagliptin phosphate
- Sitagliptin with Diet Advice (Experimental): Subjects received sitagliptin 100 mg once daily for 26 Weeks,
  and:
  Intervention on diet which includes advice on diet with a leaflet and a diary
  Interventions: Drug: sitagliptin phosphate; Behavioral: Comparator: Diet
- Sitagliptin with Diet and Physical Activity Advice (Experimental): Subjects received sitagliptin 100 mg once daily for 26 Weeks,
  and:
  Intervention on diet + physical activity which includes advice on diet and physical activity with leaflets and diaries PLUS advice on physical activity with the utilization of a pedometer: subjects were asked to walk 10,000 steps per day 5 or more days per week.
  Interventions: Drug: sitagliptin phosphate; Behavioral: Comparator: Diet; Behavioral: Comparator: Physical Activity

INTERVENTIONS:
Drug: sitagliptin phosphate — sitagliptin 100 mg once daily. Duration of treatment: 26 Weeks
Behavioral: Comparator: Diet — Diet
  Arms: Sitagliptin with Diet Advice; Sitagliptin with Diet and Physical Activity Advice
Behavioral: Comparator: Physical Activity — Physical Activity
  Arms: Sitagliptin with Diet and Physical Activity Advice

SUMMARY:
To compare the efficacy of three strategies of lifestyle changes associated with Januvia (sitagliptin) 100 mg/day in patients with Type 2 Diabetes Mellitus (T2DM) inadequately controlled by metformin (hemoglobin A1c [HbA1c] 6.5-9%). A difference between the three strategies of lifestyle changes was expected.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman aged >/= 18 years,with T2DM and treated with the maximal tolerated dose of metformin, with documented or high likely inadequate control of diabetes (HbA1c 6.5-9%)

Exclusion Criteria:

* Daily insulin treatment or one insulin dose or more within the last 8 weeks or expected insulin treatment within the next 3 months.
* Hypoglycemia unawareness or recurrent major hypoglycemia or history of acidoketosis
* Known hypersensitivity or contraindication to metformin

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1512 (Actual)
Dates: Start 2007-04-01 (Actual); Primary Completion 2009-11-19 (Actual); Study Completion 2009-11-19 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Monitor, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
http://www.merck.com/clinical-trials/pdf/Merck%20Procedure%20on%20Clinical%20Trial%20Data%20Access%20Final_Updated%20July_9_2014.pdf
  http://engagezone.msd.com/ds_documentation.php

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 1512 subjects were selected/screened, 380 subjects failed screening, leaving 1132 subjects who were randomized.
Period: Overall Study
Arm/Group | Sitagliptin With Standard of Care | Sitagliptin With Diet Advice | Sitagliptin With Diet and Physical Activity Advice
Started | 412 | 414 | 306 (306 subjects were randomized but only 305 were treated.)
Completed | 333 | 334 | 250
Not Completed | 79 | 80 | 56
Not completed — Only one reason for discontinuation | 62 | 61 | 48
Not completed — Two or more reasons for discontinuation | 17 | 19 | 8

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Sitagliptin With Standard of Care | Sitagliptin With Diet Advice | Sitagliptin With Diet and Physical Activity Advice | Total
Number analyzed (Participants) | 362 | 358 | 265 | 985
Age, Continuous [Mean (Standard Deviation); unit: years] — The Full Analysis Set (FAS) population included all selected patients with at least one measured HbA1c value after Visit 2 and having received at least one dose of sitagliptin.
  years | 58.26 (10.04) | 57.47 (9.12) | 57.30 (9.90) | 57.71 (9.68)
Sex: Female, Male [Count of Participants; unit: Participants] — The Full Analysis Set (FAS) population included all selected patients with at least one measured HbA1c value after Visit 2 and having received at least one dose of sitagliptin.
  Participants
    Female | 181 | 175 | 126 | 482
    Male | 181 | 183 | 139 | 503

OUTCOME MEASURES:

1. Primary Outcome: Hemoglobin A1c Measurement
Description: Hemoglobin A1c (HbA1c) is a measure of glycated hemoglobin in the blood. HbA1c greater than 6.5% was considered inadequately controlled.
Time Frame: Baseline and Week 24
Population: The Full Analysis Set (FAS) population included all selected patients with at least one measured HbA1c value after Visit 2 and having received at least one dose of sitagliptin. In the Standard of Care group, only 360 subjects had HbA1c Baseline evaluations.
Measure: Mean (Standard Deviation); unit: percent HbA1c
Arm/Group | Sitagliptin With Standard of Care | Sitagliptin With Diet Advice | Sitagliptin With Diet and Physical Activity Advice
Number analyzed (Participants) | 362 | 358 | 265
percent HbA1c
  Baseline (n=360, 358, and 265, respectively) | 7.37 (0.61) | 7.50 (0.66) | 7.49 (0.60)
  Week 24 (n=362, 358, and 265, respectively) | 7.33 (1.09) | 7.42 (1.15) | 7.40 (1.07)

2. Secondary Outcome: Fasting Plasma Glucose (FPG) Measurement
Description: Generally FPG values of ~5.0-7.2 mmol/L would be considered goal (American Diabetes Association).
Time Frame: Baseline and Week 24
Population: FAS population. Furthermore, only 350, 252, and 350 subjects had FPG evaluations in the Diet advice, Diet & physical activity advice, and Standard groups, respectively, at Baseline; and 303, 224, and 310 subjects had FPG evaluations in the Diet advice, Diet & physical activity advice, and Standard groups, respectively, at Week 24.
Measure: Mean (Standard Deviation); unit: mmol/L glucose
Arm/Group | Sitagliptin With Standard of Care | Sitagliptin With Diet Advice | Sitagliptin With Diet and Physical Activity Advice
Number analyzed (Participants) | 310 | 303 | 224
mmol/L glucose
  Baseline (n=350, 350, 252, respectively) | 8.87 (1.98) | 9.00 (2.03) | 8.91 (1.87)
  Week 24 (n=310, 303, and 224, respectively) | 8.21 (2.07) | 8.32 (2.08) | 8.47 (2.17)

ADVERSE EVENTS:
Time Frame: This safety data includes AEs and SAEs that occurred during treatment (Visit 2 to Visit 4).
Arm/Group | Sitagliptin With Standard of Care | Sitagliptin With Diet Advice | Sitagliptin With Diet and Physical Activity Advice
Serious Adverse Events (participants affected / at risk) | 8/412 | 18/414 | 7/305
Other Adverse Events (participants affected / at risk) | 0/412 | 0/414 | 0/305
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Sitagliptin With Standard of Care (N=412) | Sitagliptin With Diet Advice (N=414) | Sitagliptin With Diet and Physical Activity Advice (N=305)
IDIOPATHIC THROMBOCYTOPENIC PURPURA (Blood and lymphatic system disorders) | 1 (1) | 0 (0) | 0 (0)
ACUTE CORONARY SYNDROME (Cardiac disorders) | 1 (1) | 1 (1) | 0 (0)
ADAMS-STOKES SYNDROME (Cardiac disorders) | 1 (1) | 0 (0) | 0 (0)
ANGINA UNSTABLE (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MYOCARDIAL INFARCTION (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0)
MACULAR OPACITY (Eye disorders) | 0 (0) | 1 (1) | 0 (0)
INGUINAL HERNIA (Gastrointestinal disorders) | 1 (1) | 0 (0) | 0 (0)
CARDIAC DEATH (General disorders) | 0 (0) | 1 (1) | 0 (0)
SUDDEN DEATH (General disorders) | 1 (1) | 0 (0) | 0 (0)
CHOLECYSTITIS (Hepatobiliary disorders) | 0 (0) | 1 (1) | 0 (0)
ABDOMINAL WALL ABSCESS (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
EAR INFECTION (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
LARYNGITIS (Infections and infestations) | 1 (1) | 0 (0) | 0 (0)
PNEUMONIA (Infections and infestations) | 0 (0) | 1 (1) | 0 (0)
DRUG EXPOSURE DURING PREGNANCY (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1)
LIMB TRAUMATIC AMPUTATION (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
LUMBAR VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
TENDON RUPTURE (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0)
DIABETES MELLITUS (Metabolism and nutrition disorders) | 1 (1) | 0 (0) | 0 (0)
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1)
BREAST CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
FIBROMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 1 (1) | 0 (0)
LUNG NEOPLASM MALIGNANT (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1)
PROSTATE CANCER (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 2 (2)
CERVICAL ROOT PAIN (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
ENCEPHALITIS (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
SCIATICA (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1)
SYNCOPE (Nervous system disorders) | 0 (0) | 1 (1) | 0 (0)
DEPRESSION (Psychiatric disorders) | 0 (0) | 1 (1) | 0 (0)
SUICIDE ATTEMPT (Psychiatric disorders) | 1 (1) | 0 (0) | 0 (0)
RENAL NECROSIS (Renal and urinary disorders) | 0 (0) | 1 (1) | 0 (0)
GENITAL PROLAPSE (Reproductive system and breast disorders) | 0 (0) | 1 (1) | 0 (0)
PULMONARY EMBOLISM (Respiratory, thoracic and mediastinal disorders) | 1 (1) | 0 (0) | 0 (0)
RASH (Skin and subcutaneous tissue disorders) | 0 (0) | 1 (1) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Merck agreements may vary with individual investigators, but will not prohibit any investigator from publishing. Merck supports the publication of results from all centers of a multi-center trial but requests that reports based on single-site data not precede the primary publication of the entire clinical trial.